CLINICAL TRIAL: NCT05743465
Title: Evaluate the Real-World Safety Outcomes and Clinical Efficacy of Ponatinib and Other Tyrosine Kinase Inhibitors Among Chronic Myeloid Leukemia Patients
Brief Title: A Study to Evaluate Available Treatment Information of Ponatinib, Bosutinib, Imatinib, Dasatinib and Nilotinib in Adults With Chronic Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: GOR-2017-102256
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Leukemia
Keywords: Drug Therapy
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ponatinib Cohort: Participants will be classified into the cohorts based on the TKI (ponatinib, bosutinib, and others [imatinib, dasatinib, or nilotinib]) drug used on index date, stratified by prior TKI use. Participants with a ponatinib prescription identified as the index drug prior TKI use will be stratified in this cohort.
  Interventions: Other: No Intervention
- Bosutinib Cohort: Participants will be classified into the cohorts based on the TKI (ponatinib, bosutinib, and others [imatinib, dasatinib, or nilotinib]) drug used on index date, stratified by prior TKI use. Participants without ponatinib use and with bosutinib identified as the index drug prior TKI use will be stratified in this cohort.
  Interventions: Other: No Intervention
- Other TKI Cohort: Participants will be classified into the cohorts based on the TKI (ponatinib, bosutinib, and others [imatinib, dasatinib, or nilotinib]) drug used on index date, stratified by prior TKI use. Participants without ponatinib or bosutinib use and with imatinib, dasatinib, or nilotinib identified as the index drug after prior TKI use will be stratified in this cohort.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered in this study.

SUMMARY:
The aims of this study are to learn out about treatment information (including amongst others treatment patterns, safety, development of a participant's condition) ponatinib, bosutinib, imatinib, dasatinib and nilotinib using already available data. No new data will be collected from participants as part of this study and no study medicines will be provided in this study.

DETAILED DESCRIPTION:
This is a retrospective cohort analysis study in participants with chronic phase chronic myeloid leukemia (CP-CML). This study will use Humedica electronic medical record (EMR) data to evaluate the real-world treatment patterns, safety, and efficacy of ponatinib and other tyrosine kinase inhibitors (TKIs) among CP-CML participants.

The study will enroll approximately 1769 patients. Based on the TKI drug used on index date, stratified by prior TKI use, participants will be classified into the following cohorts -

* Ponatinib Cohort
* Bosutinib Cohort
* Other TKI Cohort

This is a multicenter study conducted in the United States (US). The overall duration for data collection in this trial will be approximately 5 years.

ELIGIBILITY:
Inclusion criteria:

Participants will be included in the study if they:

1. had ≥1 prescription for TKI (imatinib, dasatinib, nilotinib, bosutinib, or ponatinib) from April 1, 2013-March 31, 2017;

   * For participants with ponatinib use, the first ponatinib prescription date will be defined as the index date; for participants with bosutinib but not ponatinib use, the first bosutinib prescription date will be defined as the index date; and for participants without ponatinib and bosutinib use, the first imatinib, dasatinib, nilotinib prescription date will be defined as the index date.
   * Participants with >1 type of TKI on the index date will be dropped.
2. had ≥1 medical diagnosis for CML (International Classification of Diseases, Ninth Revision, Clinical Modification [ICD-9-CM]: 205.1; ICD-10-CM: C92.1) any time prior to the index date or within 6 months post-index date; diagnosis codes in the primary or secondary position will be used; the first CML diagnosis date will be designated as the initial CML diagnosis date;
3. were aged ≥18 years on the index date;
4. were active in the Humedica EMR data 6 months pre- and post-index date, indicated by the first and last healthcare activity in the data;

   * Participant data will be assessed until the earliest of switch to another TKI, disenrollment, death, or study end date. The minimum required duration of follow-up can be further revised based on the average duration of first-line treatment.
   * Participants who died in 6 months will be included.

Exclusion criteria:

Participants will be excluded from the study if they:

1. had ≥1 prescription for their index TKI (imatinib, dasatinib, nilotinib, bosutinib, or ponatinib) any time prior to the index date.
2. This will allow ≥6-month wash-out period, and ensure we are capturing second line participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of CP-CML and who had ≥1 prescription for TKI (imatinib, dasatinib, nilotinib, bosutinib, or ponatinib) from April 1, 2013-March 31, 2017 will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1769 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Chronic Myeloid Leukemia (CML) Participants Categorized by Sociodemographic Variables at Diagnosis | Baseline (Day 1)
  Socio-demographic variables included will include categories of Age (in years), Sex (male and female), and US geographic region.
Number of CML Participants With Baseline Clinical Characteristics of Disease Severity | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
Quan-Charlson Comorbidity Index Score | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
  The Charlson Comorbidity Index is a 19-item measure assessing comorbid conditions. The total possible score on the Charlson Comorbidity Index ranges from 0 to 37. If a condition is not present, the score for that condition is zero. The higher scores indicate greater comorbidity.
Number of CML Participants With Baseline Clinical Characteristics of Comorbidities | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
  Comorbidities will include anemia, diabetes, chronic pulmonary disease, congestive heart failure, hypertension, hypercholesterolemia, obesity, renal disease, moderate to severe liver disease, dementia, acquired immune deficiency syndrome (AIDS)/human immunodeficiency virus (HIV).
Number of CML Participants With Baseline Clinical Characteristics of Concomitant Medication | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
  Concomitant medication will include antithrombotic agents (anticoagulants, antiplatelet), antihypertensive, and antidiabetic drugs (angiotensin converting enzyme inhibitor, angiotensin receptor blocker, beta blockers and statins) and antidiabetic drugs (metformin, sulfonylurea, thiazolidinedione, insulin and other antidiabetic drugs).
Number of Previous Treatments of Tyrosine Kinase Inhibitors (TKI) Drugs in Participants with CML | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
  The number of TKI drugs used prior to the index date will be identified. The type of the 1^st and 2^nd TKI drugs will be identified.
Duration Between Last TKI Run-out Date to the Index Date for Participants with CML | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
  Time from the run-out date of the last prescription to the index date will be calculated. If the run-out date passed the index date, the gap will be counted as 0.
Number of Participants with Bone Marrow Stem Cell Transplant | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
Clinical Characteristics Assessed by Number of Participants With Major Adverse Cardiac Events (MACE), Arterial Occlusive Events (AOEs), and Venous Thrombotic Events (VTEs) | Up to 6 months prior to the day of initiation of TKI drug i.e., Day 1
  MACE will be categorized as myocardial infarction and stroke. AOE will be categorized according to cardiovascular events, cerebrovascular events and peripheral vascular arterial events will be categorized as pulmonary embolism (PE) and deep vein thrombosis (DVT).
Treatment Patterns Based on Duration of Index Treatment | Up to approximately 5 years
  Time from the first prescription of the index drug to the run-out date of the last prescription of the index drug, or 1 day before a new TKI prescription date, whichever occurred earlier.

SECONDARY OUTCOMES:
Number of Participants With BCR-ABL and Bone Marrow Testing | Up to approximately 5 years
  BCR-ABL test will include participants tested for BCR-ABL mutation, such as T315I, and participants with a diagnostic marrow test.
Treatment Patterns Based on Mean Starting Daily Dose and Average Daily Dose in Participants with CML | Up to approximately 5 years
  The mean daily and average dose of the first prescription in the treatment line will be calculated. The starting and average daily dose will be classified as low, standard, and high for each drug cohort.
Number of CML Participants With Disease Severity as per Medstat Disease Staging Clinical Criteria Version 5.21 | Up to approximately 5 years
  The disease severity will include categories of low, moderate, and high severity.
Treatment Patterns Based on Number of Participants With CML on Concomitant Medication | Up to approximately 5 years
  The concomitant medications will include antithrombotic agents (anticoagulants, antiplatelet), antihypertensive, and antidiabetic drugs.
Number of Participants With CML With Treatment-Free Gap of the Index Treatment | Up to approximately 5 years
Disease Progression | Up to approximately 5 years
  Disease progression will be defined as having a change of disease severity from low severity in the baseline period to moderate or high severity in the current line, or from moderate severity in the baseline period to high severity in the current line OR a change in TKI type, addition of chemotherapy agents, or allogeneic stem cell transplant procedure OR mortality.
Percentage of CML Participants With Complications | Up to approximately 5 years
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the interval between the first does of study treatment and death due to any cause, censored at the last contact date when the participant was alive.
Progression Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time in days from the index date to the first observed disease progression.
Number of Participants with Atleast one Adverse Event, Major Adverse Cardiac Event (MACE), Arterial Occlusive Events (AOEs) and Venous Thrombotic Events (VTEs) | Up to approximately 5 years
  AE is any untoward medical occurrence in participant administered medicinal investigational drug. Untoward medical occurrence does not necessarily have to have causal relationship with the treatment. MACE will be categorized as myocardial infarction and stroke. AOE will be categorized according to cardiovascular events, cerebrovascular events and peripheral vascular arterial events will be categorized as PE and DVT.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5a2b267658b5473c?idFilter=%5B%22GOR-2017-102256%22%5D